CLINICAL TRIAL: NCT04864496
Title: Effects of Oral N- Acetylcysteine on Macular Function in Retinitis Pigmentosa; a Phase 2 Randomized Controlled Trial
Brief Title: Effects of Treatment With N- Acetylcysteine on Visual Outcomes in Patients With Retinitis Pigmentosa
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1400
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prescribe N-acetylcysteine tablets (Active Comparator)
  Interventions: Drug: Prescribe N-acetylcysteine tablets
- Prescribe placebo tablets (Placebo Comparator)
  Interventions: Drug: Prescribe placebo tablets

INTERVENTIONS:
Drug: Prescribe N-acetylcysteine tablets — N-acetylcysteine tablets ,1200 mg two times daily
  Arms: Prescribe N-acetylcysteine tablets
Drug: Prescribe placebo tablets — manufactured by Daroo Salamat Pharmed, two times daily
  Arms: Prescribe placebo tablets

SUMMARY:
Retinitis pigmentosa (RP) is an inherited retinal disease with great heterogeneity. RP comprises a large group of genetic disorders causing progressive loss of vision. Despite many suggested treatments, there is actually no effective therapy for most types of RP at present. Mutations that cause RP initially lead to rod cell death. After rod photoreceptors' death, cone photoreceptors also gradually die. There are several hypotheses as to why mutation-induced rod photoreceptor cell death invariably leads to gradual dysfunction and death of cone photoreceptors resulting in severe visual acuity loss and blindness. Rods constitute 95 percent of cells in the outer retina. As they degenerate, oxygen consumption is reduced and the level of tissue oxygen markedly increases. After rods degeneration, several markers of oxidative damage appear in cones. This oxidative stress over time may lead to cone dysfunction and death. Antioxidants reduce markers of oxidative damage and promote cone function and survival. In RP, cone death occurs as a result of the death of rods, rather than as the result of the pathogenic mutations and therefore treatment with antioxidants may have the potential to be applied to all patients with RP irrespective of the disease-causing mutation.

N-acetylcysteine is a derivative of L cysteine that plays a role in the biosynthesis of glutathione and neutralizes reactive oxygen species. It also has a direct antioxidant activity via its reactive sulfhydryl agent. Its systemic use shows an acceptable safety profile. It has been shown that the use of systemic N-acetylcysteine provides significant intraocular concentration and antioxidant activity that may lead to the promotion of cone function and survival.

In a recent phase 1 randomized clinical trial (RCT), it was revealed that oral N-acetylcysteine (NAC) was safe and well-tolerated in patients with moderately advanced RP and might improve sub-optimally functioning macular cones. The authors concluded that a randomized, placebo-controlled trial is needed to determine if oral NAC can provide long-term stabilization and/or improvement in visual function in patients with RP. In this phase 2 RCT, eligible patients with the diagnosis of moderately advanced RP are randomly divided into two groups; treatment group (N-acetylcysteine tablets) and controls (placebo). Each group will be treated for 6 months. In this study, we will investigate if the use of oral N- acetylcysteine as a potent antioxidant agent can slow down or reverse the disease process in RP patients with prior moderate loss of vision. It may potentially demonstrate a treatment modality regardless of the genetic type of RP. The primary outcome measure will be the stability or improvement of the best-corrected visual acuity (BCVA). The secondary outcome measures will be changes in color vision, electroretinogram, visual field, structural OCT indices after 6 months. The same parameters will be re-evaluated 3 months after discontinuation of treatment at month 9.

ELIGIBILITY:
Inclusion Criteria:

* RP patients with the best-corrected visual acuity (BCVA) between 20/30 and 20/120.

Exclusion Criteria:

* Patients with other types of retinal dystrophy
* Systemic or syndromic RP
* RP patients with cystoid macular edema (CME) and the presence of cystoid changes in the foveal area
* RP patients with other concomitant ocular diseases
* RP patients with a history of any ocular surgery or intravitreal injection within 6 months before the study enrollment
* RP patients who have received any supplemental drugs during the past three months before the study enrollment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-17 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Change of the best corrected visual acuity (BCVA) from baseline to month 6 | 6 months
  ETDRS chart

SECONDARY OUTCOMES:
Change of the ellipsoid zone (EZ) width from baseline to month 6 | 6 months
  spectral domain optical coherence tomography (SD-OCT)
Changes of the wave amplitude of the flicker response from baseline to month 6 | 6 months
  Full field electroretinograph (ffERG) testing
Change of the foveal and macular sensitivity from baseline to month 6 | 6 months
  visual field testing
Change of the color discrimination parameters from baseline to month 6 | 6 months
  D15 Fransworth 100 Hue Test

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran